CLINICAL TRIAL: NCT00840762
Title: A Randomized Comparison of Virco®TYPE HIV-1 Testing Versus Expert Interpretation of Genotypic Results for Control of HIV-1 Replication
Brief Title: A Comparison of Virco®TYPE HIV-1 Testing Versus Expert Interpretation of Genotypic Results for Control of HIV-1 Replication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruth M. Rothstein CORE Center (Other)
Collaborators: Virco (Industry)
Responsible Party: David E. Barker, MD, The Ruth M. Rothstein CORE Center of Cook County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 07-118
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV-1; HIV; HIV Genotypic testing; resistance
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VircoType HIV-1 (Experimental): Genotypic HIV resistance testing results interpreted by VircoType HIV-1 algorithm
  Interventions: Other: VircoType HIV-1 genotypic interpretation
- Local Expert review (Active Comparator): Local Expert HIV genotypic review, as per Badri, S. et al CID 2003
  Interventions: Other: Local Expert Review of HIV Genotypic resistance testing

INTERVENTIONS:
Other: VircoType HIV-1 genotypic interpretation — VircoType HIV-1 genotypic interpretation
  Arms: VircoType HIV-1
Other: Local Expert Review of HIV Genotypic resistance testing — Local Expert Review of HIV Genotypic resistance testing
  Arms: Local Expert review

SUMMARY:
The investigators seek to determine whether Virco®TYPE HIV-1 provides benefits equivalent to those provided by local expert review. The investigators propose that clinic patients of the Ruth M. Rothstein CORE Center who are having genotypic testing performed will be randomized in a 1:1 fashion to local expert review and to Virco®TYPE HIV-1. Results of either method will be shared with primary HIV care providers. Patient outcomes will be reviewed at a time point equal to or greater than 2 months and 6 months following the change in antiretroviral medications following the testing

DETAILED DESCRIPTION:
Patients having some documented genotypic HIV resistance but having more than one fully active medication will be randomized to either local review or algorithmic review by VircoType HIV-1.

ELIGIBILITY:
Inclusion Criteria:

* HIV resistance testing that demonstrates resistance to at least one drug
* Patients of the CORE Center, Chicago Illinois

Exclusion Criteria:

* Wild type HIV on resistance testing or less than or equal to one active antiretroviral medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with viral load <1000 60days after HIV regimen change | 60 days
Proportion of patients with viral load <1000 180 days after HIV regimen change | 180 days

SECONDARY OUTCOMES:
Proportion of patients with undetectable viral load 60days after HIV regimen change | 60 days
Proportion of patients with undetectable viral load 180days after HIV regimen change | 180 days
CD4 Cell count change in each arm at 60 and 180 days | 60 and 180 days
Proportion of patients whose regimen fails and who require repeat resistance testing at 180 and 360 days | 180 and 360 days
Comparison of number of active drugs predicted by each review method and number of actual active drugs prescribed | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: David E Barker, MD, Principal Investigator — Ruth M. Rothstein CORE Center
Locations (1):
- The Ruth M. Rothstein CORE Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Badri SM, Adeyemi OM, Max BE, Zagorski BM, Barker DE. How does expert advice impact genotypic resistance testing in clinical practice? Clin Infect Dis. 2003 Sep 1;37(5):708-13. doi: 10.1086/377266. Epub 2003 Aug 15. PMID 12942405
- See also: The CORE Center — http://www.corecenter.org/
- See also: Cook County Hospital Department of Medicine — http://www.cchil.org/index.html
- See also: UIC College of Pharmacy — http://www.uic.edu/pharmacy/about_the_college/index.php